CLINICAL TRIAL: NCT00040443
Title: Efficacy And Safety Of CX516 (900 mg t.i.d.) In Elderly Participants With Mild Cognitive Impairment. A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group 4-week Study.
Brief Title: Efficacy And Safety Of CX516 In Elderly Participants With Mild Cognitive Impairment.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RespireRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORX-CX516-012.1
Record Dates: First submitted 2002-06-26; First posted 2002-06-28 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Memory Loss; Alzheimer's Disease; Brain Aging; Ampalex®; CX516
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Alzheimer Disease | interventions — 1-(quinoxalin-6-ylcarbonyl)piperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CX516 (Experimental): CX516 - 900 mg
  Interventions: Drug: CX516
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CX516
  Arms: CX516
Drug: Placebo
  Arms: Placebo

SUMMARY:
Glutamate is fundamentally involved in learning and memory. Memory loss associated with mild cognitive impairment may be due to loss of glutamate receptors in the aging brain. There is evidence CX516 enhances brain activity by specifically targeting remaining glutamate receptors in the affected portions of the brain. This study will test the safety and efficacy of CX516 in the symptomatic treatment of participants with mild cognitive impairment.

ELIGIBILITY:
Inclusion criteria

* Clinical diagnosis of mild cognitive impairment
* Good general health with no additional diseases that would interfere with the study.

Exclusion criteria

* Any significant neurologic disease (other than suspected incipient Alzheimer's disease), such as Parkinson's disease, stroke, TIA's, multi-infarct dementia, Huntington's disease, head trauma, chronic CNS infection.
* History of major depression or another major psychiatric disorder within the past 6 months.
* History of schizophrenia, mania or recurrent psychotic episodes.
* History of alcohol or DSM IV-diagnosed substance abuse or dependence disorder within the past year.
* History of blackout, epilepsy or seizures, or an abnormal EEG as judged by the Investigator and considering the age of the participant.
* Any clinically significant hepatic, renal, cardiovascular, pulmonary, gastrointestinal or hematological illness or unstable medical condition which could interfere with drug safety, or absorption, distribution, metabolism and excretion, or lead to difficulty complying with the protocol.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2002-04; Primary Completion 2003-08 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Pivotal Research Centers, Peoria, Arizona
  - University of California Irvine, Irvine, California
  - University of California at Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Sun Coast Gerontology Center, University of South Florida, Tampa, Florida
  - Mercy Mayo Clinic, Des Moines, Iowa
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CX516: CX516 - 900 mg
  CX516 (Ampalex®)
- Placebo: Placebo to CX516 900 mg
  CX516 (Ampalex®)
Period: Overall Study
Arm/Group | CX516 | Placebo
Started | 84 | 91
Completed | 84 | 91
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CX516 | Placebo | Total
Number analyzed (Participants) | 84 | 91 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (7.7) | 70.3 (8.5) | 71.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 47 | 53 | 100

OUTCOME MEASURES:

1. Primary Outcome: 15-Item Word List Delayed Recall
Description: The 15-Item Word List delayed recall score is used as a clinical measure of episodic memory, and was the primary outcome variable for this study. Episodic memory of the type addressed by delayed recall of lists and stories (i.e., in the WMS-R logical memory tests and 15-item World List recall tests) is among the earliest deficits during aging and MCI compared to other aspects of cognition (attention, reaction time, language, etc). It was decided to use the 15-item Word List delayed recall test as the primary outcome measure due to its sensitivity in the assessment of MCI.
  The possible score range for the 15-item Word List Delayed Recall test is 0 to 15. A clinical improvement of MCI or dementia would be characterized by an increase in the score due to an increase in the number of words recalled.
Time Frame: 28 Days
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale - change from baseline
Groups:
- CX516: CX516 - 900 mg (3 X 300 mg)
  CX516 (Ampalex®)
- Placebo: Placebo to CX516 300 mg
  CX516 (Ampalex®)
Arm/Group | CX516 | Placebo
Number analyzed (Participants) | 84 | 91
units on a scale - change from baseline | -0.3 (2.3) | -0.5 (2.3)
Statistical Analysis 1: Comparison: CX516 vs Placebo; Test type: Other; p < .05, t-test, 2 sided; Mean Difference (Final Values) = 5, Standard Error of Mean 1

ADVERSE EVENTS:
Time Frame: 28 Day treatment 8 week followup
Arm/Group | CX516 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/91
Serious Adverse Events (participants affected / at risk) | 3/84 | 1/91
Other Adverse Events (participants affected / at risk) | 68/84 | 56/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CX516 (N=84) | Placebo (N=91)
neutrophil count decrease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
moderate urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CX516 (N=84) | Placebo (N=91)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 6 (6) | 4 (4)
Urinary Tract Infections (Infections and infestations) | 3 (3) | 0 (0)
Creatinin increased (Investigations) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 12 (12) | 3 (3)
Insominia (Psychiatric disorders) | 7 (7) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhea NOS (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 14 (14) | 2 (2)
Eructation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Flatulance (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 17 (17) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Neutrophil decreased (Investigations) | 6 (6) | 3 (3)
back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 25 (25) | 17 (17)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No